CLINICAL TRIAL: NCT06177340
Title: Visualization by the Nanoscope System During Sacrospinofixation
Brief Title: Nanoscope System During Sacrospinofixation
Acronym: SF-CAM
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5408
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Sacrospinofixation
Keywords: Nanoscope system; sacrospinofixation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacrospinofixation: patient who benefited from anterior and/or posterior sacrospinofixation using the Nanoscope system
  Interventions: Device: visualization of the sacrospinous ligament

INTERVENTIONS:
Device: visualization of the sacrospinous ligament — visualization of the sacrospinous ligament by the Nanoscope system during sacrospinofixation

SUMMARY:
Sacrospinofixation is one of the reference techniques for the treatment of vaginal prolapse. It consists of fixing a non-absorbable thread on the sacrosciatic ligament unilaterally or bilaterally to correct a urogenital prolapse.

The technical difficulty is linked to the fact that the approach to the sacrosciatic ligament is palpatory without visual control. However, if the thread is not well fixed in the ligament, there is a risk of this suture coming loose and therefore of recurrence of the prolapse. On the other hand, due to the vascular and nervous proximity (pudendal nerve), vascular complications such as hemorrhage and/or hematoma have been described by vascular lesion during the passage of the needle through this ligament. Nervous complications due to pinning of the pudendal nerve or its nerve branches have also been described, which can cause after-effects of pain or even chronic dyspareunia.

Clearly and precisely visualizing the sacrosciatic ligament and the vascular and nervous structures with a microcamera could make it possible to better correct the prolapse and limit recurrences, but also to avoid these serious and disabling complications.

The Nanoscope system, which can be used in routine practice as part of sacrospinofixation, could make it possible to obtain visibility of tissues under vision control. Thus the precise visualization of the sacrospinous ligament would allow an easier approach and therefore more precise surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* patient who benefited from anterior and/or posterior sacrospinofixation using the nanoscope system
* person having expressed his non-opposition

Exclusion Criteria:

* inability to understand the information given
* person deprived of liberty
* person under guardianship

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study concerns patients who underwent anterior and/or posterior sacrospinofixation surgery to correct a prolapse and for whom the Nanoscope system was used.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
visualization of the sacrospinous ligament | during surgery
  Obtaining visualization of the sacrospinous ligament by the Nanoscope system during sacrospinofixation (binary criterion: yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Lyon, France

IPD SHARING:
Plan to Share IPD: No